CLINICAL TRIAL: NCT04419714
Title: A Single Center, Single Arm, Quantitative Study Assessing Performance of TatchSleep as a Tool to Aid in Sleep Apnea Analysis
Brief Title: TatchSleep as a Tool to Aid in Sleep Apnea Analysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wesper Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: TCH-103
Record Dates: First submitted 2020-06-03; First posted 2020-06-05 (Actual); Results first posted 2025-08-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-07

CONDITIONS: Sleep Apnea; Sleep Disorder
MeSH Terms: conditions — Sleep Apnea Syndromes; Sleep Wake Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- TatchSleep Pro Test Arm (Experimental): This is the only arm tested in the study. Individuals within this arm were male and female participants, that were at least 18 years or older. Every participant wore the TatchSleep Pro device while simultaneously undergoing an in-lab PSG.
  Interventions: Device: TatchSleep

INTERVENTIONS:
Device: TatchSleep — Wearable measurement device

SUMMARY:
This is a single center, single-arm, quantitative study evaluating the efficacy of the TatchSleep wireless sensor patches as a tool to aid in sleep apnea analysis as compared to an overnight PSG evaluation.

DETAILED DESCRIPTION:
This is a multi-center, single-arm, quantitative study evaluating the effectiveness of the TatchSleep Pro wireless sensors as a tool to aid in sleep apnea diagnosis as compared to an overnight PSG evaluation.

Investigators will identify approximately 50 eligible patients who have been recommended to receive an overnight PSG for the detection/evaluation of sleep apnea. After informed consent is obtained, a brief sleep-related medical history will be collected including relevant demographics. Females of childbearing potential will be asked to undergo a urine dipstick pregnancy test to determine their eligibility for inclusion in the study.

Patients will undergo their PSG test while simultaneously wearing 2 TatchSleep Pro patches and an FDA-cleared pulse oximeter compatible with and connected to the TatchSleep Pro system for a single night at the clinic. The same make and model of pulse oximeter will be used for all subjects. Patients will be observed overnight by trained sleep technicians who will setup the TatchSleep Pro device and collect the sleep data via the companion smartphone application.

A follow-up communication will be made with patients within 5 days after the sleep study to assess any adverse events. Following the data collection, sleep data from PSG and TatchSleep Pro will be scored by an independent qualified sleep technologist (the primary reader) to yield an analysis of the accuracy of TatchSleep Pro compared with the PSG signals. At least one and up to two additional readers (secondary readers) will score only the TatchSleep Pro data to obtain an estimate of inter-rater reliability.

ELIGIBILITY:
Inclusion Criteria:

1. Be at least 18 years of age
2. Have a referral to the clinical site from a physician, to complete an overnight polysomnogram test for sleep apnea detection or follow-up.
3. Be able to read, write, and speak English
4. Be willing and able to wear 3 TatchSleep patches, in conjunction with a polysomnogram, for a single night.
5. The patient must be able to sign a written informed consent form prior to the initiation of any study procedures. Adult patients unable to provide written informed consent on their own behalf will not be eligible for the study.

Exclusion Criteria:

1. Latex allergy
2. Morbidly obese patients (BMI>39.5)
3. Females who are pregnant, trying to get pregnant or who have a urine test positive for pregnancy on the day of the study
4. Women who are breast-feeding
5. Any known health condition that, in the opinion of the Investigator, would exclude the patient from participating in the study.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2021-06-10 (Actual); Primary Completion 2021-11-04 (Actual); Study Completion 2021-11-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Imran M Ahmed, MD, Principal Investigator — ontefiore Medical Center; Suzanne Pearson, RPSGT, RST, Principal Investigator — The Valley Hospital Center for Sleep Medicine; Matthew L Uhles, RPSGT, RST, Principal Investigator — Clayton Sleep Institute
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Sleep Apnea Measurement Device (Test Arm): There is only one arm of this study. The arm includes adults that used the TatchSleep Pro device, which is a medical device that detects and measures sleep apnea.
Period: Overall Study
Arm/Group | Sleep Apnea Measurement Device (Test Arm)
Started | 53
Completed | 45
Not Completed | 8
Not completed — Technical Fault | 5
Not completed — Protocol Deviation | 2
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Males and females, 18 years of age or older. Measure Analysis Population Description: Overall tested population was 53 but protocol deviation, equipment errors, and one withdrawal lead to 45 being analyzed
Arm/Group | TatchSleep Pro Test Arm
Number analyzed (Participants) | 45
Age, Categorical [Count of Participants; unit: Participants] — Population: Overall tested population was 53 but protocol deviation, equipment errors, and one withdrawal lead to 45 being analyzed
  Participants
    <=18 years | 0
    Between 18 and 65 years | 32
    >=65 years | 13
Age, Continuous [Mean (Full Range); unit: years] | 48.8 [21 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8
  Not Hispanic or Latino | 37
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 10
  White | 26
  More than one race | 1
  Unknown or Not Reported | 6
Region of Enrollment [Number; unit: participants]
  United States | 45

OUTCOME MEASURES:

1. Primary Outcome: Correlation Between Polysomnography (PSG) and Tatch Apnea/Hypopnea Index (AHI)
Description: The correlation between AHI (3% desaturation criterion) measured by the TatchSleep Pro device and in-lab PSG will be assessed. Agreement between the two modalities will be analyzed using Bland-Altman analysis, and Pearson correlation coefficients will be calculated for AHI and ODI (3%). This outcome evaluates the concordance between TatchSleep Pro and PSG for key respiratory indices.
Time Frame: 12 hours
Population: Subjects that used TatchSleep Pro while simultaneously undergoing a Polysomnography (PSG) sleep study
Measure: Number (95% Confidence Interval); unit: correlation coefficient (r)
Arm/Group | TatchSleep Pro Test Arm
Number analyzed (Participants) | 45
correlation coefficient (r) | 0.95 [0.92 to 0.97]

2. Secondary Outcome: Percent Agreement of AHI Severity Classification Between TatchSleep Pro and Polysomnography
Description: Agreement in AHI severity classification (Normal, Mild, Moderate, Severe) between TatchSleep Pro and in-lab PSG was assessed using blinded scoring. Severity assignments from both devices were compared using percent agreement.
Time Frame: 12 hours
Population: Participants that simultaneously wore the TatchSleep Pro while undergoing a Polysomnography (PSG) sleep study
Measure: Number; unit: Percent Agreement
Groups:
- Medical Device TatchSleep Pro: Test Arm: Participants that simultaneously wore the TatchSleep Pro while undergoing a Polysomnography (PSG) sleep study
Arm/Group | Medical Device TatchSleep Pro: Test Arm
Number analyzed (Participants) | 45
Percent Agreement | 89

3. Secondary Outcome: Agreement Between TatchSleep Pro and PSG on AHI Severity Using Cohen's Kappa
Description: Agreement in AHI severity classification (Normal, Mild, Moderate, Severe) between TatchSleep Pro and in-lab PSG was assessed using blinded scorers. The level of agreement was quantified using the weighted Cohen's kappa coefficient.
Time Frame: 12 hours
Population: Participants that simultaneously wore the TatchSleep Pro while undergoing a Polysomnography (PSG) sleep study
Measure: Number (95% Confidence Interval); unit: kappa
Arm/Group | Medical Device TatchSleep Pro: Test Arm
Number analyzed (Participants) | 45
kappa | 0.82 [0.70 to 0.94]

ADVERSE EVENTS:
Time Frame: 2 days
Description: Adverse event data were collected using a systematic assessment approach. Participants were monitored throughout the 2-day study period, and any adverse events were recorded via structured interviews and observation by study staff.
Groups:
- Medical Device: TatchSleep Pro: Single Arm: Participants that wore the TatchSleep Pro while simultaneously undergoing a Polysomnography (PSG) sleep study
Arm/Group | Medical Device: TatchSleep Pro: Single Arm
All-Cause Mortality (participants affected / at risk) | 0/45
Serious Adverse Events (participants affected / at risk) | 0/45
Other Adverse Events (participants affected / at risk) | 0/45

LIMITATIONS AND CAVEATS:
This study was conducted at a single site with a relatively small sample size (n = 45), which may limit generalizability

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-04-26): https://cdn.clinicaltrials.gov/large-docs/14/NCT04419714/Prot_SAP_000.pdf
  • Informed Consent Form (2021-04-28): https://cdn.clinicaltrials.gov/large-docs/14/NCT04419714/ICF_001.pdf